CLINICAL TRIAL: NCT00377741
Title: Relative Bioavailability Study of Ganciclovir From the Pro-drug, Valganciclovir, in Lung Transplant Recipients With or Without Cystic Fibrosis
Brief Title: A Relative Bioavailability Study of Valcyte (Valganciclovir) in Lung Transplant Recipients With or Without Cystic Fibrosis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WP18046
Record Dates: First submitted 2006-09-15; First posted 2006-09-18 (Estimated); Results first posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-11

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: valganciclovir [Valcyte]

INTERVENTIONS:
Drug: valganciclovir [Valcyte] — 900mg po

SUMMARY:
This study will assess the relative bioavailability of ganciclovir from the pro-drug valganciclovir in lung transplant recipients with or without cystic fibrosis. Each patient will receive 900mg valganciclovir daily for the period specified at their center, starting as soon as possible after the transplant. Pharmacokinetic assessments will be made provided that steady-state kinetics of ganciclovir and immunosuppressive drugs have been obtained (>=4 days of drug therapy). Blood samples for pharmacokinetic analysis will be taken up to 24h post-dose on one occasion. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients, >=14 years of age;
* first lung or heart-lung transplant recipient;
* at risk of CMV disease (D+R-,D+R+ or D-R+);
* estimated creatinine clearance >=60mL/min;
* stable immunosuppressive and 900mg Valcyte dosing regimens (>=4 days) prior to pharmacokinetic assessments.

Exclusion Criteria:

* history of any adverse reaction to acyclovir, valacyclovir, ganciclovir or valganciclovir;
* evidence of graft rejection;
* patient has received anti-CMV prophylaxis with a treatment other than cytogam, ganciclovir or valganciclovir between transplant and screening.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2004-12; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (5):
  - Los Angeles, California
  - Denver, Colorado
  - Durham, North Carolina
  - Cleveland, Ohio
  - Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 31 participants were included from 5 centers in the United States of America. This study was conducted between 01 December 2004 and 30 June 2006.
Pre-assignment Details: Participants were received 900 mg of commercial medication of valganciclovir tablet daily for >= 4 days prior to study Day 1 so as to achieve steady-state kinetics of ganciclovir.
Groups:
- Cystic Fibrosis (CF): Participants with cystic fibrosis (CF) received a single oral dose of valganciclovir 900 mg
- Non-Cystic Fibrosis (Non-CF): Participants with non-cystic fibrosis (Non-CF) received a single oral dose of valganciclovir 900 mg
Period: Overall Study
Arm/Group | Cystic Fibrosis (CF) | Non-Cystic Fibrosis (Non-CF)
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cystic Fibrosis (CF) | Non-Cystic Fibrosis (Non-CF) | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.8 (9.82) | 51.6 (8.66) | 40.4 (14.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 6 | 10 | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under The Observed Plasma Concentration-Time Curve Between Dosing Intervals AUC(0-tau)
Description: The area under the plasma concentration-time curve from time zero to end of dosing interval (AUC [0-tau]) is a measure of the plasma ganciclovir concentration from time zero to end of dosing interval. It was computed using the linear trapezoidal rule. The pharmacokinetic parameters of valganciclovir were measured in plasma of all participants following a single oral dose valganciclovir at 900 mg on Day 1.
Time Frame: Pre-dose, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12 and 24 hours post-dose
Population: The Pharmacokinetic (PK) analysis population included all participants who received study medication and had at least one PK sample.
Measure: Mean (Standard Deviation); unit: h*mcg/mL
Arm/Group | Cystic Fibrosis (CF) | Non-Cystic Fibrosis (Non-CF)
Number analyzed (Participants) | 16 | 15
h*mcg/mL | 66.2 (31.3) | 54.1 (16.6)
Statistical Analysis 1: Comparison: Cystic Fibrosis (CF) vs Non-Cystic Fibrosis (Non-CF); Test type: Superiority or Other; Mean exposure ratio for AUC(0-tau) = 1.24, 90% CI 2-sided [0.98 to 1.55]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ganciclovir
Description: The Cmax is defined as maximum observed Ganciclovir concentration. Cmax of valganciclovir were measured in plasma of all participants following a single tablet dose Valganciclovir at 900 mg at start of treatment on Day 1.
Time Frame: Pre-dose, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12 and 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Cystic Fibrosis (CF) | Non-Cystic Fibrosis (Non-CF)
Number analyzed (Participants) | 16 | 15
μg/mL | 8.46 (3.16) | 7.54 (2.23)
Statistical Analysis 1: Comparison: Cystic Fibrosis (CF) vs Non-Cystic Fibrosis (Non-CF); Test type: Superiority or Other; Mean exposure ratio for Cmax = 1.12, 90% CI 2-sided [0.88 to 1.42]

3. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Ganciclovir
Description: The Tmax is defined as time to reach maximum observed Ganciclovir concentration. The pharmacokinetic parameters of Valganciclovir were measured in plasma of all participants following a single tablet dose Valganciclovir at 900 mg at start of treatment on Day 1.
Time Frame: Pre-dose, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12 and 24 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Cystic Fibrosis (CF) | Non-Cystic Fibrosis (Non-CF)
Number analyzed (Participants) | 16 | 15
h | 1.99 [1.00 to 4.07] | 1.98 [0.92 to 5.97]

4. Secondary Outcome: Apparent Elimination Rate (Kelim) of Ganciclovir
Description: The apparent elimination rate is equal to the magnitude of the slope from the log-linear regression of plasma concentration versus time over the interval t to 24, where t is the first time-point used for this regression. Kelim was not reported for those participants for whom R-squared (adjusted) was lower than 0.70.
Time Frame: Pre-dose, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12 and 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Cystic Fibrosis (CF) | Non-Cystic Fibrosis (Non-CF)
Number analyzed (Participants) | 16 | 15
1/h | 4.43 (0.745) | 4.91 (0.684)

5. Secondary Outcome: Plasma Half-Life (T1/2) of Ganciclovir
Description: Plasma half-life is the time measured for the plasma concentration to decrease by one half. The pharmacokinetic parameters of Valganciclovir were measured in plasma of all participants following a single tablet dose Valganciclovir at 900 mg at start of treatment on Day 1. T1/2 was not reported for those participants for whom R-squared (adjusted) was lower than 0.70.
Time Frame: Pre-dose, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12 and 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cystic Fibrosis (CF) | Non-Cystic Fibrosis (Non-CF)
Number analyzed (Participants) | 16 | 15
h | 4.43 (0.75) | 4.91 (0.68)

ADVERSE EVENTS:
Time Frame: Up to 4 Weeks
Description: Serious adverse events (SAEs) and non-serious AEs were reported for the safety population which included all patients who were enrolled on the study and had at least one safety assessment, whether withdrawn prematurely or no were included in the safety analysis.
Arm/Group | Cystic Fibrosis (CF) | Non-Cystic Fibrosis (Non-CF)
Serious Adverse Events (participants affected / at risk) | 3/16 | 1/16
Other Adverse Events (participants affected / at risk) | 5/16 | 4/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cystic Fibrosis (CF) (N=16) | Non-Cystic Fibrosis (Non-CF) (N=16)
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Chills (General disorders) | 1 | 0
Enterococcal Bacteraemia (Infections and infestations) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cystic Fibrosis (CF) (N=16) | Non-Cystic Fibrosis (Non-CF) (N=15)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Fatigue (General disorders) | 0 | 1
Transplant Rejection (Immune system disorders) | 1 | 0
Pulmonary Function Test Decreased (Investigations) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.